CLINICAL TRIAL: NCT02724163
Title: International Randomised Phase III Clinical Trial in Children With Acute Myeloid Leukaemia - Incorporating an Embedded Dose Finding Study for Gemtuzumab Ozogamicin in Combination With Induction Chemotherapy
Brief Title: International Randomised Phase III Clinical Trial in Children With Acute Myeloid Leukaemia
Acronym: Myechild01
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other); Cancer Research UK (Other); National Cancer Institute, France (Other Government); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RG_14-088; 2014-005066-30 (EudraCT Number)
Record Dates: First submitted 2016-01-08; First posted 2016-03-31 (Estimated); Last update posted 2021-10-08 (Actual); Status verified 2021-09

CONDITIONS: Acute Myeloid Leukaemia
Keywords: Acute Myeloid Leukaemia; Children; Gemtuzumab ozogamicin; Liposomal daunorubicin; Mitoxantrone; Randomised controlled trial; Risk stratification; Minimal residual disease; Stem cell transplant
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Neoplasm, Residual | interventions — Gemtuzumab; Daunorubicin; Mitoxantrone; fludarabine; Cytarabine; Busulfan; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Mitoxantrone (Active Comparator): Course 1
  * Mitoxantrone: 12 mg/m2 daily by IV infusion over 1 hour on days 1, 2, 3 and 4 (total 4 doses).
  * Cytarabine:100 mg/m2 12 hourly by IV bolus on days 1-10 inclusive (total 20 doses).
  Course 2
  * Mitoxantrone: 12 mg/m2 daily by IV infusion over 1 hour on days 1, 2 and 3 (total 3 doses).
  * Cytarabine: 100 mg/m2 12 hourly by IV bolus on days 1-8 inclusive (total 16 doses).
  Interventions: Drug: Mitoxantrone; Drug: Cytarabine
- Liposomal daunorubicin (Experimental): Randomisation 1 (R1)) closed early to recruitment on 8th September 2017, due to liposomal daunorubicin manufacturing issues resulting in unavailability of the drug.
  Course 1
  * Liposomal daunorubicin: 80 mg/m2 daily by 1 hour IV infusion on days 1, 3 and 5 (total 3 doses).
  * Cytarabine: 100 mg/m2 12 hourly by IV bolus on days 1-10 inclusive (total 20 doses).
  Course 2
  * Liposomal daunorubicin: 60 mg/m2 daily by 1 hour IV infusion on days 1, 3 and 5 (total 3 doses).
  * Cytarabine: 100 mg/m2 12 hourly by IV bolus on days 1-8 inclusive (total 16 doses).
  Interventions: Drug: Liposomal daunorubicin; Drug: Cytarabine
- Gemtuzumab Ozogamicin Dose Finding Study (Experimental): * Cohort 1: 1x3mg/m2 IV infusion over 2hours on day 4.
  * Cohort 2: 2x3mg/m2 IV infusion over 2hours on day 4 and day 7.
  * Cohort 3: 3x3mg/m2 IV infusion over 2hours on days 4, 7 and 10.
  Interventions: Drug: Gemtuzumab ozogamicin
- High dose cytarabine (Active Comparator): Two courses of Cytarabine: 3 g/m2 12 hourly by IV infusion over 4 hours on days 1, 3 and 5 (total 6 doses).
  Interventions: Drug: Cytarabine
- Fludarabine & cytarabine (Experimental): Two courses of:
  * Fludarabine: 30 mg/m2 daily by IV infusion over 30 minutes on days 1-5 inclusive (total 5 doses).
  * Cytarabine: 2 g/m2 daily by IV infusion over 4 hours on days 1-5 inclusive (total 5 doses).The cytarabine infusion should be started 4 hours after the start of the fludarabine infusion
  Interventions: Drug: Fludarabine; Drug: Cytarabine
- Myeloablative conditioning (Active Comparator): * Busulfan Area Under the Curve (AUC) 70-100mg/L x hr by IV infusion over 3 hours, given 12 hourly on days -10 to -7 (8 doses).
  * Cyclophosphamide 50mg/kg/day by IV infusion over 1 hour, on days -5 to -2 (4 doses).
  Interventions: Drug: Busulfan; Drug: Cyclophosphamide
- Reduced intensity conditioning (Experimental): * Busulfan AUC60-65mg/L X hr by IV infusion over 3 hours, given 12 hourly on days -5 to -2 (8 doses).
  * Fludarabine 30mg/m2/day by IV infusion over 30 minutes on days -8 to -3 (6 doses).
  Interventions: Drug: Fludarabine; Drug: Busulfan

INTERVENTIONS:
Drug: Gemtuzumab ozogamicin — Antibody-conjugated chemotherapy agent.
  Other Names: Mylotarg
  Arms: Gemtuzumab Ozogamicin Dose Finding Study
Drug: Liposomal daunorubicin — Anthracycline
  (Randomisation 1 (R1)) closed early to recruitment on 8th September 2017, due to liposomal daunorubicin manufacturing issues resulting in unavailability of the drug.
  Arms: Liposomal daunorubicin
Drug: Mitoxantrone — DNA-reactive agent
  Arms: Mitoxantrone
Drug: Fludarabine — A water-soluble fluorinated nucleotide analogue of the antiviral agent vidarabine.
  Arms: Fludarabine & cytarabine; Reduced intensity conditioning
Drug: Cytarabine — Pyrimidine nucleoside analogue, an antineoplastic agent.
  Arms: Fludarabine & cytarabine; High dose cytarabine; Liposomal daunorubicin; Mitoxantrone
Drug: Busulfan — Alkylsulfonate
  Arms: Myeloablative conditioning; Reduced intensity conditioning
Drug: Cyclophosphamide — A nitrogen mustard alkylating agent from the oxazaphosphorine group
  Arms: Myeloablative conditioning

SUMMARY:
The main purpose of this study is :

1. To establish which number of doses of gemtuzumab ozogamicin (up to a maximum of 3 doses) is tolerated and can be safety delivered in combination with cytarabine plus mitoxantrone or liposomal daunorubicin in induction
2. To compare mitoxantrone (anthracenedione) & cytarabine with liposomal daunorubicin (anthracycline) & cytarabine as induction therapy. (Randomisation 1 (R1) closed early to recruitment on 8th September 2017, due to liposomal daunorubicin manufacturing issues resulting in unavailability of the drug.)
3. To compare a single dose of gemtuzumab ozogamicin with the optimum tolerated number of doses of gemtuzumab ozogamicin (identified by the dose-finding study) when combined with induction chemotherapy.
4. To compare two consolidation regimens: high dose cytarabine (HD Ara-C) and fludarabine & cytarabine (FLA) in standard risk patients.
5. To compare the toxicity and effectiveness of two haemopoietic stem cell transplant (HSCT) conditioning regimens of different intensity: conventional myeloablative conditioning (MAC) with busulfan/cyclophosphamide and reduced intensity conditioning (RIC) with fludarabine/busulfan.

DETAILED DESCRIPTION:
MyeChild 01 is an international phase III clinical trial in children with acute myeloid leukaemia (AML); a disease with significant mortality. It will compare two induction chemotherapy regimens: mitoxantrone and cytarabine (current standard treatment) with liposomal daunorubicin and cytarabine. This will test liposomal daunorubicin, which is believed to be less cardiotoxic than similar conventional drugs, although this is unproven. (Randomisation 1 (R1) closed early to recruitment on 8th September 2017, due to liposomal daunorubicin manufacturing issues resulting in unavailability of the drug.)

Patients responding well to induction chemotherapy are eligible for a randomisation of two consolidation regimens: high dose cytarabine (current standard treatment) or fludarabine and cytarabine (FLA); a regimen commonly used in patients with relapsed disease, testing whether FLA is more effective in front line therapy than standard consolidation treatment. Patients with cytogenetic features associated with a higher risk of relapse and those responding sub-optimally to induction treatment are candidates for haemopoietic stem cell transplant (HSCT) and are eligible for a randomisation comparing two HSCT conditioning regimens: myeloablative conditioning (MAC) (current UNited Kingdom (UK) standard) or reduced intensity conditioning (RIC). HSCT has not consistently shown benefit in high risk patients because the mortality associated with the procedure has outweighed the advantage from a reduction in relapse risk. This will test whether reducing the intensity of conditioning improves survival by reducing transplant related deaths without increasing the relapse rate. The trial incorporates a dose finding study for gemtuzumab ozogamicin. The aim is to identify the optimum tolerated number of doses of gemtuzumab ozogamicin (up to a total of 3 doses), which can be safely combined with either of the induction chemotherapy regimens and then to compare this number of doses with one dose of gemtuzumab ozogamicin. The intensity of treatment will be directed by cytogenetics/molecular genetics and response assessed by minimal residual disease (MRD) levels measured by flow cytometry and molecular methodology.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for trial entry

* Diagnosis of acute myeloid leukaemia (AML) /high risk Myelodysplastic syndrome (MDS) (>10% blasts in the bone marrow)/isolated myeloid sarcoma (MS) (either de novo or secondary).
* Age <18 years at trial entry.
* No prior chemotherapy or biological therapy for AML/high risk MDS/isolated MS other than that permitted in the protocol.
* Normal cardiac function defined as fractional shortening ≥28% or ejection fraction ≥55%.
* Fit for protocol chemotherapy.
* Documented negative pregnancy test for female patients of childbearing potential.
* Patient agrees to use effective contraception (patients of child bearing potential).
* Written informed consent from the patient and/or parent/legal guardian.

Inclusion criteria for participation in the gemtuzumab ozogamicin dose finding study:

Centres must be formally activated in order to be take part in the embedded dose escalation study. Please contact the trial office for further information.

* Patient meets the inclusion criteria for trial entry.
* Age:

  * ≥12 months for the major dose finding study
  * ≥ 12 weeks and <12 months for the minor dose finding study
* Normal renal function defined as calculated creatinine clearance ≥90ml/min/1.73m2.
* Normal hepatic function defined as total bilirubin ≤2.5 upper limit of normal (ULN) for age unless it is caused by leukaemic involvement or Gilbert's syndrome or similar disorder.
* Alanine transaminase (ALT) or aspartate transaminase (AST) ≤10 x ULN for age.
* Written informed consent from the patient and/or parent/legal guardian.

Inclusion criteria for treatment with gemtuzumab ozogamicin for patients not participating in the gemtuzumab ozogamicin dose finding study or R2.

* Patient meets the inclusion criteria for trial entry (section 4.1.1)
* Age:

  * ≥12 months
  * ≥ 12 weeks
  * ≥28 days and <12 weeks (patients will receive a maximum of one dose of gemtuzumab ozogamicin)
* Normal renal function, defined as calculated creatinine clearance ≥90 ml/min/1.73m2
* Normal hepatic function, defined as total bilirubin ≤2.5 upper limit of normal (ULN) for age and not due to leukaemic involvement or Gilbert's syndrome or similar disorder
* ALT or AST ≤10 x ULN for age
* Written informed consent from the patient and/or parent/legal guardian

Inclusion criteria for participation in R2.(once open to randomisation in the applicable age group)

• Patient meets the inclusion criteria for trial entry

Patient age:

* ≥12 months
* ≥12 weeks (once R2 open in patients aged ≥12 weeks and <12 months)
* Normal renal function defined as calculated creatinine clearance ≥90ml/min/1.73m2.
* Normal hepatic function defined as total bilirubin ≤2.5 ULN for age and not due to leukaemic involvement or Gilbert's syndrome or similar disorder.
* ALT or AST ≤10 x ULN for age.
* Written informed consent from the patient and/or parent/legal guardian.

Inclusion criteria for participation in R3.

* Patient meets the inclusion criteria for trial entry
* Induction treatment as per MyeChild 01 protocol or treated with 2 courses of mitoxantrone & cytarabine off trial.
* Minimal residual disease (MRD) response (performed in MyeChild 01 centralised laboratories, see national MyeChild 01 Laboratory Manual):

  * Patients with good risk cytogenetics/molecular genetics and a MRD level <0.1% by flow after course 2, or a decrease in transcript levels of >3 logs after course 2 for those with an informative molecular marker, but without an informative marker of sufficient sensitivity for flow MRD monitoring or
  * Patients with intermediate risk cytogenetics/molecular genetics with a MRD level <0.1% by flow after course 1 and course 2, or a decrease in transcript levels of >3 logs after course 1 and course 2 for those with an informative molecular marker, but without an informative marker of sufficient sensitivity for flow MRD monitoring.
* Written informed consent from the patient and/or parent/legal guardian.

Inclusion criteria for participation in R4.

* Patient meets the inclusion criteria for trial entry
* Induction treatment as per MyeChild 01 protocol or treated with 1 or 2 courses of mitoxantrone & cytarabine ± treatment intensification with fludarabine, cytarabine & idarubicin (FLA-Ida) off trial.
* Patient is in complete remission (CR) or CR with incomplete blood count recovery (CRi) defined as <5% blasts confirmed by flow cytometry/ molecular/FISH in a bone marrow aspirate taken within 6 weeks prior to randomisation to R4.
* Patient meets one of the following criteria and is a candidate for HSCT as per the protocol:

  * High risk after course 1 (all patients with poor risk cytogenetics and patients with intermediate risk cytogenetics who fail to achieve CR/CRi).
  * Intermediate risk cytogenetics with MRD >0.1% after course 1 and 2 measured by flow. If no flow MRD marker of sufficient sensitivity is identified, a molecular MRD marker with a sensitivity of >0.1% may be used.
  * Good risk cytogenetics with flow MRD >0.1% confirmed by a decrease in molecular MRD of <3 logs or rising transcript levels after course 3 despite treatment intensification (FLA-Ida) and after discussion with the Clinical Co-ordinators.
* Availability of a 9-10/10 human leukocyte antigen (HLA) matched family or unrelated donor or 5-8/8 matched cord blood unit with an adequate cell dose as defined by the protocol section 17.1.
* Written informed consent from the patient and/or parent/legal guardian.

Exclusion Criteria:

Exclusion criteria for all randomisations

* Acute Promyelocytic Leukaemia.
* Myeloid Leukaemia of Down Syndrome.
* Blast crisis of chronic myeloid leukaemia.
* Relapsed or refractory AML.
* Bone marrow failure syndromes.
* Prior anthracycline exposure which would inhibit the delivery of study anthracyclines.
* Concurrent treatment or administration of any other experimental drug or with any other biological therapy for AML/high risk MDS/isolated MS.
* Pregnant or lactating females.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 700 (Estimated)
Dates: Start 2016-04 (Actual); Primary Completion 2031-12 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLTs). | Incidence of DLTs will be evaluated up to day 45 post course 1 and course 2 of induction chemotherapy.
Event Free Survival (EFS). | Event free survival (EFS) will be evaluated as the time from randomisation one to the first event, up to 16 years.
  The primary analysis will be carried out once the last patient has a minimum of 1 year follow up. EFS estimates will be presented at 24 months along with 95% confidence intervals.
Event Free Survival (EFS). | Event free survival (EFS) will be evaluated as the time from randomisation two to the first event, up to 16 years..
  The primary analysis will be carried out once the last patient has a minimum of 1 year follow up. EFS estimates will be presented at 24 months along with 95% confidence intervals.
Relapse free survival (RFS). | Relapse free survival (RFS) will be evaluated as the time of randomisation three to the first relapse or death from any cause, up to 16 years.
  The primary analysis will be carried out once the last patient has a minimum of 1 year follow up. RFS estimates will be presented at 24 months along with 95% confidence intervals.
Early treatment related adverse reactions. | Early treatment related adverse reactions will be evaluated at day 100 post-transplant.
  Early treatment related adverse reactions defined as the incidence by day 100 post-transplant of grade 3-5 toxicity for the following systems using the National Cancer Institute (NCI) Common Terminology Criteria v4:
  * Cardiac (pericardial effusion/Left ventricular systolic dysfunction).
  * Respiratory, thoracic and mediastinal (hypoxia/pneumonitis).
  * Gastrointestinal (GI) (diarrhoea/typhlitis/upper and lower GI haemorrhage).
  * Investigations (bilirubin).
  * Renal and Urinary (acute kidney injury/haematuria).
  * Nervous system (seizure).
Relapse free survival (RFS). | Relapse free survival (RFS) will be evaluated as the time of randomisation four to the first relapse or death from any cause, up to 16 years.
  The primary analysis will be carried out once the last patient has a minimum of 1 year follow up. RFS estimates will be presented at 12 months along with 95% confidence intervals.

SECONDARY OUTCOMES:
The nature, incidence and severity of adverse events (AEs) (gemtuzumab ozogamicin dose finding study). | Evaluated by day 45 post course 1 and course 2.
Response measured by bone marrow assessment using morphology and minimal residual disease (MRD) assessment (gemtuzumab ozogamicin dose finding study). | Evaluated by day 45 post course 1 and course 2.
  Response is assessed by morphology confirmed by MRD levels measured by flow cytometry, molecular methods or fluorescence in situ hybridisation (FISH) as defined in the protocol, in combination with platelet and neutrophil counts. These results of these assessments will be combined to determine the patient's disease response using the response criteria defined in the protocol.
Serum pharmacokinetic (PK) parameters of gemtuzumab ozogamicin: Clearance (CL) (gemtuzumab ozogamicin dose finding study) | Evaluated up to one month after the first dose of gemtuzumab ozogamicin.
  Serum PK parameters will be measured using serial samples taken at multiple timepoints during course 1 and at 1 month post first dose of gemtuzumab ozogamicin as defined in the protocol by dose cohort.
Serum pharmacokinetic (PK) parameters of gemtuzumab ozogamicin: Volume of distribution (Vd) (gemtuzumab ozogamicin dose finding study) | Evaluated up to one month after the first dose of gemtuzumab ozogamicin.
  Serum PK parameters will be measured using serial samples taken at multiple timepoints during course 1 and at 1 month post first dose of gemtuzumab ozogamicin as defined in the protocol by dose cohort.
Complete remission (CR) (R1 & R2). | Evaluated and presented at the completion of course 1 and 2 of treatment up to a maximum of 45 days post each course of treatment
  Evaluated using remission status at completion of course 1 and course 2.
Reasons for failure to achieve CR (R1 & R2). | Evaluated and presented at the completion of course 1 and 2 of treatment, up to a maximum of 45 days post each course of treatment.
  Evaluated as resistant disease, induction death or not evaluable.This will be evaluated at completion of course 1 and 2 of treatment, once patient's blood counts have recovered or reason for non-recovery has been determined.
Cumulative Incidence of Relapse (CIR) (all randomisations). | Evaluated as time from randomisation to the relevant question to relapse, up to 16 years.
  The primary analysis will be carried out once the last patient has a minimum of 1 year follow up. CIR estimates will be presented at 24 months along with 95% confidence intervals for randomisations 1, 2 and 3, and at 12 months for randomisation 4.
Death in CR (DCR) (R1, R2 & R3). | Evaluated as time from randomisation to relevant question to date of death from any cause in patients who have achieved CR, up to 16 years.
  The primary analysis will be carried out once the last patient has a minimum of 1 year follow up. DCR estimates will be presented at 24 months along with 95% confidence intervals.
Event Free Survival (EFS) (R1, R2 & R3). | Evaluated as time from randomisation to the relevant question to the first of failure to achieve CR (recorded as an event on day 1), relapse, secondary malignancy or death from any cause, up to 16 years.
  The primary analysis will be carried out once the last patient has a minimum of 1 year follow up. EFS estimates will be presented at 24 months along with 95% confidence intervals.
Overall Survival (OS) (all randomisations). | Evaluated as time from randomisation to the relevant question to death from any cause or date last seen for patients who are alive at the end of the trial, up to 16 years.
  The primary analysis will be carried out once the last patient has a minimum of 1 year follow up. OS estimates will be presented at 24 months along with 95% confidence intervals for randomisations 1, 2 and 3, and at 12 months for randomisation 4.
Incidence of toxicities (all randomisations). | Evaluated 30 days after end of trial treatment.
Incidence of cardiotoxicity (R1, R2 & R4 only). | Evaluated 30 days after end of trial treatment.
Incidence of bilirubin of grade 3 of higher (R2 & R4 only). | Evaluated 30 days after end of trial treatment.
Incidence of Veno-Occlusive Disease (R2 & R4 only). | Evaluated 30 days after end of trial treatment.
Minimal Residual Disease (MRD) clearance after course 1 & 2 (R1 & R2 only). | Evaluated and presented at completion of course 1 and 2 of treatment, up to a maximum of 45 days post each course of treatment.
  Evaluated using MRD result at completion of course 1 and 2 once patient's blood counts have recovered or reason for non-recovery has been determined.
Time to haematological recovery (all randomisations). | Evaluated by day 45 post course 1 and course 2.
  Evaluated using the date of haematological recovery (platelets to >=80 x 10^9/L, and neutrophils to >=1.0 x 10^9/L). The primary analysis will be carried out once the last patient has a minimum of 1 year follow up. Time to haematological recovery estimates will be presented at 45 days post course 1 and course 2 of treatment along with 95% confidence intervals.
Days in hospital after each course of treatment (all randomisations). | Evaluated once all patients have completed trial treatment.
  Total number of days spent in hospital for each course of treatment, collected from date of randomisation until count recovery after final course of treatment, up to a maximum of 45 days post the final course of treatment. This will be summarised per course of treatment.
Incidence of mixed chimerism at day 100 post-transplant (R4 only). | Evaluated at day 100 post-transplant.
Treatment Related Mortality (TRM) (R4 only). | Evaluated as time in days between randomisation to R4 and death which is unrelated to the underlying disease and considered related to the transplant procedure.
  The primary analysis will be carried out once the last patient has a minimum of 1 year follow up which is estimated to be 7 years after the start of recruitment. TRM estimates will be presented at 12 months along with 95% confidence intervals.
Gonadal function (R4 only). | Evaluated at 1 year post-transplant and at the end of follow-up, which is estimated to be through to study completion, an average timeframe of 10 years.
  The method of assessment will be by scale (Tanner scale) and physiological parameters. This will be evaluated at 1 year post-transplant and at the end of study follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Brenda Gibson, Principal Investigator — Royal Hospital for Children Glasgow
Locations (68):
- Australia (8):
  - Women and Children's Hospital Adelaide, Adelaide
  - Queensland Children's Hospital, Brisbane
  - Monash Children's Hospital, Melbourne
  - Royal Childrens Hospital, Melbourne
  - John Hunter Children's Hopsital, New Lambton Heights
  - Perth Children's Hospital, Perth
  - Sydney Children's Hospital, Sydney
  - The Childrens Hospital At Westmead, Westmead
- France (28):
  - Centre Hospitalier Universitaire Amiens - Picardie, Amiens
  - Centre Hospitalier Universitaire D'angers, Angers
  - Centre Hospitalier Regional Universitaire Besancon - Hopital Jean Minjoz, Besançon
  - Centre Hospitalier Universitaire De Bordeaux - Hopital Pellegrin, Bordeaux
  - Centre Hospitalier Regional Universitaire Brest - Hopital Morvan, Brest
  - Centre Hospitalier Universitaire De Caen, Caen
  - Centre Hospitalier Universitaire De Clermont-ferrand, Clermont-Ferrand
  - Centre Hospitalier Universitaire Dijon Bourgogne - Hopital D'enfants, Dijon
  - Centre Hospitalier Universitaire De Grenoble, Grenoble
  - Hopital Jeanne Dr Flandre, Lille
  - Centre Hospitalier Universitaire De Limoges, Limoges
  - Centre Leon Berard, Lyon
  - Hopital De La Timone, Marseille
  - Centre Hospitalier Regional Universitaire Montpellier - Hopital Arnaud-de-villeneuve, Montpellier
  - Centre Hospitalier Universitaire De Nancy, Nancy
  - Centre Hospitalier Universitaire De Nantes, Nantes
  - Centre Hospitalier Universitaire De NICE, Nice
  - Hopital Armand Trousseau, Paris
  - Hopital Robert Debre, Paris
  - Hopital Saint Louis, Paris
  - Centre Hospitalier Universitaire De Poitiers, Poitiers
  - Chu De Reims, Reims
  - Centre Hospitalier Universitaire De Rennes - Hopital Sud, Rennes
  - Centre Hospitalier Universitaire De Rouen, Rouen
  - Centre Hospitalier Universitaire Saint-etienne, Saint-Etienne
  - Strasbourg Hautepierre, Strasbourg
  - Centre Hospitalier Universitaire De Toulouse - Hopital Des Enfants, Toulouse
  - Centre Hospitalier Regional Universitaire De Tours - Hopital Clocheville, Tours
- Our Lady's Hospital for Sick Children, Dublin, Ireland
- New Zealand (2):
  - Starship Childrens Hospital, Auckland
  - Christchurch Hospital, Christchurch
- Switzerland (9):
  - Kantonsspital Aarau, Aarau
  - Universitäts-Kinderspital beider, Basel
  - Ospedale San Giovanni, Bellinzona
  - Inselspital Bern, Bern
  - Hug Hopitaux Universitaires De Geneve, Geneva
  - Centre Hospitalier Universitaire Vaudois Chuv Lausanne, Lausanne
  - Luzerner Kantonspital - Kinderspital Luzern, Lucerne
  - Ostschweizer Kinderspital, Sankt Gallen
  - University Children's Hospital Zurich, Zurich
- United Kingdom (20):
  - Royal Belfast Hospital for Sick Children, Belfast, County Antrim
  - Royal Aberdeen Children's Hospital, Aberdeen
  - Aberdeen Royal Infirmary, NHS Grampian, Aberdeen
  - Birmingham Children's Hospital NHS Foundation Trust, Birmingham
  - University Hospitals Bristol NHS Foundation Trust, Bristol
  - Addenbrookes Hospital, Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Cardiff and Vale University Health Board, Noah's Ark Children's Hospital for Wales, Cardiff
  - NHS Lothian, Royal Hospital for Sick Children, Edinburgh
  - NHS Greater Glasgow and Clyde, The Royal Hospital for Children, Glasgow
  - Leeds General Infirmary, Leeds Teaching Hospitals NHS Trust, Leeds
  - Alder Hey Children's NHS Foundation Trust, Liverpool
  - University College London Hospitals NHS Foundation Trust, London
  - The Royal Marsden NHS Foundation Trust, London
  - Great Ormond Street Hospital For Children NHS Trust, London
  - Royal Manchester Childrens' Hospital , Central Manchester University Hospitals NHS Foundation Trust, Manchester
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust, Newcastle
  - Nottingham University Hospitals NHS Trust, Nottingham
  - John Radcliffe Hospital, Oxford Radcliffe Hospitals NHS Trust, Oxford
  - Sheffield Children's NHS Foundation Trust, Sheffield
  - Southampton University Hospitals NHS Trust, Southampton

IPD SHARING:
Plan to Share IPD: No